CLINICAL TRIAL: NCT03899363
Title: A Prospective, Randomized Controlled Trial of Two Treatment for a Mallet Finger of Tendinous Origin
Brief Title: Two Treatment for a Mallet Finger of Tendinous Origin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2018-08-417
Record Dates: First submitted 2019-03-19; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Mallet Finger
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery (Experimental)
  Interventions: Procedure: custom thermoplastic orthosis
- custom thermoplastic orthosis (Active Comparator)
  Interventions: Procedure: custom thermoplastic orthosis

INTERVENTIONS:
Procedure: custom thermoplastic orthosis — extended the DIP by a custom thermoplastic orthosis or the Kirschner wire through the joint
  Other Names: Kirschner wire

SUMMARY:
A randomized clinical trial, with patients treated either by a custom thermoplastic orthosis or by the Kirschner wire with the distal interphalangeal (DIP) joint extended.

Evaluating the treatment efficacy of the operation management compared with a conventional orthosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a mallet finger, with or without fracture;
* Age≥18 years

Exclusion Criteria:

* Open lesions
* Mallet fractures with subluxation of the DIP
* Delays in treatment >2 weeks
* DM
* RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion(ROM) of the DIP joint from the first week up to the 16th week after the treatment completed | The first visit(Enrolled and completed treatment), 8 weeks after first visit(two weeks after 6 weeks fixation), 16 weeks(4 weeks after six weeks Rehabilitation)
  Use a Protractor to measure the maximum degree of active flexion of the DIP joint at the first visit and at the end treatment; Use a Protractor to measure the maximum degree of active extension of the DIP joint at the start of immobilization and end of treatment.
  (If the maximum degree of active flexion of two time periods are 40° and 40°，respectively; the maximum degree of active extension of two time periods are 20° and -10°，respectively. We could get the range of motion of the DIP joint of two time periods are 20°~40° and -10°~40°，respectively. The maximum extension angle increased by 30 degrees).To assess whether there was a statistical difference in ROM changes between the two groups before and after treatment.

IPD SHARING:
Plan to Share IPD: No